CLINICAL TRIAL: NCT03870841
Title: An Open-label Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Inhaled PC945 in Adult Cystic Fibrosis (CF) Patients With Persistent Pulmonary Aspergillus Fumigatus Infection
Brief Title: The Effect of PC945 on Aspergillus Fumigatus Lung Infection in Patients With Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is being terminated early as a result of the coronavirus (COVID-19) outbreak.
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC_ASP_003; 2018-000243-87 (EudraCT Number)
Record Dates: First submitted 2018-10-24; First posted 2019-03-12 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Aspergillosis; Cystic Fibrosis
MeSH Terms: conditions — Aspergillosis; Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PC945 (Experimental): PC945 5mg once daily
  Interventions: Drug: PC945

INTERVENTIONS:
Drug: PC945 — PC945, nebulized

SUMMARY:
This study tests the effects of an experimental drug PC945 in people with cystic fibrosis whose lungs are infected by the fungus Aspergillus fumigatus.

PC945 may be useful in treating patients infected with Aspergillus fumigatus as, unlike the usual treatments, it is inhaled into the lung and has been designed to stay there and treat the infection. Participants will continue to be treated with their usual cystic fibrosis treatment and will also receive PC945. The amount of fungus in the patients' phlegm will be measured over the course of the study. The study will take place at multiple sites in UK and will include approximately 18 participants. The maximum study duration will be about 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be male or female, aged 18 years inclusive or older (at the time of consent).
2. Subject must be willing and able to adhere to the restrictions and prohibitions required by this protocol.
3. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose and requirements of the study and that they are willing to participate.
4. A confirmed diagnosis of CF by standard criteria.
5. Subject is able to produce sputum.
6. A history of persistently positive A. fumigatus sputum cultures from at least 2 sputum samples in the last year, the most recent of which must have been within the last 6 months.
7. Subject must have a positive sputum fungal culture at screening with one or more colonies of A. fumigatus detected using a modified standard approach.

Exclusion Criteria:

1. Any other disease or condition, which in the Investigator's medical opinion would preclude the subject's participation in a clinical trial.
2. Is taking inhaled amphotericin B or has taken it within 7 weeks of Day 1.
3. Is taking systemic steroid treatment or has taken it within 4 weeks of Day 1. Subjects considered to be stable on a systemic steroid dose of <15 mg for at least a month will not be excluded.
4. Is taking systemic antifungal treatment (intravenous, oral or inhaled) or has received antifungal therapy (intravenous, oral or inhaled) within 6 weeks of Day 1.
5. If female, the subject is pregnant (e.g., has a positive serum β human chorionic gonadotropin (β-hCG) at screening or a positive urinary pregnancy test pre-dose on Day 1), lactating or breast feeding.
6. Any respiratory exacerbation within 2 weeks of the start of the study.
7. Any upper respiratory tract infection or signs or symptoms thereof within 2 weeks prior to dosing.
8. Positive culture for Mycobacterium abscessus within 12 months before screening or between screening and baseline, or currently receiving treatment for Mycobacterium abscessus.
9. Has chronic, active hepatitis or a positive hepatitis B surface antigen or positive hepatitis C antibody result at screening.
10. Is taking antiretroviral protease inhibitor therapy.
11. Allergy to any of the active or inactive ingredients in the study medication.
12. History of drug (or other) allergy or intolerance that, in the opinion of the Investigator or Pulmocide Medical Monitor, would contraindicate their participation.
13. Clinically significant haemoptysis (>200 mL per episode) within 90 days before screening.
14. Subject is mentally or legally incapacitated. 19 July 2018 CONFIDENTIAL Page 27 of 58 Pulmocide Ltd Clinical Protocol PC_ASP_003
15. Subject is employed or is a first-degree relative of anyone employed by Pulmocide, a participating clinical trial site, or any contract research organisation involved in the study.
16. Any other reason that the Investigator considers makes the subject unsuitable to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Baseline to Day 84
Proportion of participants who meet the markedly abnormal criteria for 12-lead ECG assessment at lease once post dose | Baseline to Day 84
Proportion of participants who meet the markedly abnormal criteria for safety laboratory assessment at lease once post dose | Baseline to Day 84
Proportion of participants who meet the markedly abnormal criteria for vital signs assessment at lease once post dose | Baseline to Day 84
Predicted post bronchodilator forced expiratory volume in 1 second (FEV1) values | Baseline to Day 84
Forced vital capacity (FVC) values | Baseline to Day 84
Peak expiratory flow rate values (PEFR) | Baseline to Day 84
Maximum expiratory flow values (MEF25-75) | Baseline to Day 84
Breathlessness visual analogue scale rating, change over time | Baseline to Day 84
  Symptom severity rated from "Best ever" to "Worst possible"
Cough visual analogue scale rating, change over time | Baseline to Day 84
  Symptom severity rated from "Best ever" to "Worst possible"
Area under the curve from time 0 to 2 h post-dose (AUC0-2) | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
Maximum plasma concentration | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
Concentration at the end of the dosage interval (Ctrough) | Baseline to Day 84
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable

SECONDARY OUTCOMES:
Change in the number of sputum A. fumigatus colony forming units (CFU) | Baseline to Day 84
A. fumigatus status (presence or absence) in subjects with a baseline A. fumigatus-positive sputum culture | Day 1 to Day 84
Change in sputum A. fumigatus measured by quantitative polymerase chain reaction (qPCR) | Baseline to Day 84
Change in the serum concentration of A. fumigatus-specific immunoglobulins G (IgG) | Baseline to Day 84
Change in serum Total immunoglobulin E (IgE) levels | Baseline to Day 84
Change in serum Aspergillus-specific IgE levels | Baseline to Day 84
Correlation between A. fumigatus measured by qPCR and clinical response | Baseline to Day 84
Cystic Fibrosis Questionnaire - Revised (CFQ-R) score | Baseline to Day 84
Sputum consistency, including presence of blood | Baseline to Day 84
  Categorical variable
Sputum colour | Baseline to Day 84
  Categorical variable using standardised colour chart.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - Northwest Lung Research Centre, Manchester